CLINICAL TRIAL: NCT00355485
Title: Microdermabrasion for Acne Vulgaris
Brief Title: Microdermabrasion for Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Darius J. Karimipour, M.D., Clinical Assistant Professor, University of Michigan Department of Dermatology
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Derm 563
Record Dates: First submitted 2006-07-21; First posted 2006-07-24 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Acne Vulgaris
Keywords: Acne; Microdermabrasion
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Microdermabrasion Treatment (Experimental): Bilateral, split-face comparison in which one half of the face will be randomly assigned to receive the microdermabrasion treatment(s) while the other half of the face will not. Subjects will receive a series of microdermabrasion treatment sessions (up to 6) spaced one to two weeks apart. In all cases, microdermabrasion treatment parameters will be within those accepted in cosmetic work.
  Interventions: Device: microdermabrasion

INTERVENTIONS:
Device: microdermabrasion — Device: Bellamed microdermabrasion system produced by Bella products or the Altair Diamondtome System.
  Subjects will receive a series of microdermabrasion treatment sessions (up to 6) spaced one to two weeks apart.

SUMMARY:
The purpose of this research project is to study the effect of micordermabrasion to try to improve the appearance of facial acne. The microdermabrasion machine is a hand-held device that directs pressurized aluminum oxide crystals at its target accompanied by a suction device. It is not yet clear how much improvement can be seen with these treatments or exactly how the skin's response causes these improvements. In this study, we are interested in learning how well microdermabrasion works to improve the symptoms of acne.

DETAILED DESCRIPTION:
Acne vulgaris remains among the most common cutaneous disorders, impacting the vast majority of people at some point during their lives. It is associated with significant psychosocial morbidity, and there remains the need for efficacious and low risk therapeutic options.

Microdermabrasion is a technique combining abrasion and negative pressure used primarily in the treatment of aging skin. It has also been proposed to improve acne presumably through a comedolytic effect. Negative pressure and abrasion may remove debris from follicular orifices that act as a nidus for acne lesions. Many physicians and spas use micordermabrasion as a treatment for acne, however, there has never been a randomized controlled trial to substantiate this practice.

We propose to evaluate the efficacy of microdermabrasion in the treatment of inflammatory acne. We will use the Bellamed microdermabrasion system produced by Bella products or the Altair Diamondtome System.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 years or older of either gender and of any racial/ethnic group.
* Presence of clinically evident acne vulgaris of the facial skin.
* Subjects must be in generally good health.
* Subjects must be able and willing to comply with the requirements of the protocol.
* Subjects must live within a reasonable driving distance of Ann Arbor, Michigan, and/or be able to attend all of the scheduled appointments during the study.

Exclusion Criteria:

* Oral retinoid use within 6 months of entry into the study.
* Systemic acne therapies (oral antibiotics) within 4 weeks of entry into the study.
* Topical acne therapies (retinoids,antibiotics) within 2 weeks of entry into the study.
* Laser or superficial chemical peels at the sites to be treated within 3 months of entry into the study.
* Subjects with a history of dermabrasion or laser resurfacing at the sites to be treated.
* Use of topical lipid absorbing substances (Clinac AC) within 2 weeks of entry into the study.
* Non-compliant subjects.
* Subjects with a significant medical history or concurrent illness/condition which the investigator(s) feel is not safe for study participation.
* Subjects using alcohol-based topical solutions or "exfoliating" agents within 2 weeks of entry into the study.
* Subjects with a history of very frequent herpes simplex infections of the face or with clinical evidence of active herpes simplex infections.
* Pregnant or nursing females.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Counts of specific types of acne lesions. | These lesions will be counted at baseline, at follow-up evaluation visits during the treatment series, and every 1-4 weeks following the final treatment for a total of up to 18 weeks.

SECONDARY OUTCOMES:
Clinical photographs | Photographs may be obtained at baseline, at follow-up evaluation visits during the treatment series, and every 1-4 weeks following the final treatment for a total of up to 18 weeks.
Subject self-assessment questionnaire | At end of treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: John J Voorhees, MD, Study Chair — University of Michigan; Darius Karimipour, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States